CLINICAL TRIAL: NCT02166294
Title: A Multi-center, Randomized, Parallel, Crossover Design Study of Non-healing Diabetic Foot Ulcers, Treated With Cryopreserved, Umbilical Cord Allograft (NEOX® CORD 1K) Versus Standard of Care That Are Followed for 12 Weeks
Brief Title: NEOX® CORD 1K vs Standard of Care in Non-healing Diabetic Foot Ulcers
Acronym: CONDUCT I
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Amniox Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NE-2001
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Foot Ulcer, Diabetic
Keywords: Foot; Ulcer; Diabetes; Amputation; Limb salvage
MeSH Terms: conditions — Diabetic Foot; Ulcer; Diabetes Mellitus | interventions — Cryopreservation; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- NEOX® CORD 1K (Experimental): Cryopreserved, umbilical cord allograft (NEOX® CORD 1K) with off-loading instructions.
  Interventions: Other: NEOX® CORD 1K
- Pressure bandage (Active Comparator): Standard of Care Pressure bandage with off-loading instructions
  Interventions: Procedure: Standard of Care (Pressure Bandage)
- Standard of Care Cross over to NEOX (Experimental): Subjects in the Standard of Care (pressure bandage) group that have not healed greater than 50% at the Week 12 visit, or have a wound that is worsening, will be offered participation in the cross-over arm of the trial. The cross-over arm of the study will be treated with NEOX CORD 1K and followed for 12 weeks.
  Interventions: Other: NEOX® CORD 1K; Procedure: Standard of Care (Pressure Bandage)

INTERVENTIONS:
Other: NEOX® CORD 1K — Amniotic Membrane Tissue is fetal membrane tissue that comprises the innermost layer of the human placenta, and the outermost lining of the umbilical cord. In addition to amniotic membrane, the umbilical cord also contains Wharton's jelly, a rich source of proteoglycans and growth factors. These tissues share the same cell origin as the fetus and serve to protect the fetus during development. This product does not contain live cells.
  Other Names: cryopreserved, umbilical cord allograft; cryopreserved human amniotic membrane and umbilical cord; c-hAMUC; AM/UC
  Arms: NEOX® CORD 1K; Standard of Care Cross over to NEOX
Procedure: Standard of Care (Pressure Bandage) — Standard of Care wound, pressure dressing applied as needed at each visit.
  Arms: Pressure bandage; Standard of Care Cross over to NEOX

SUMMARY:
In this randomized, multi-center, cross-over study, the efficacy and safety of NEOX® CORD 1K will be evaluated in patients suffering from non-healing diabetic foot ulcers. NEOX® CORD 1K is a cryopreserved human Amniotic Membrane and Umbilical Cord (AM/UC) matrix intended for use as a wound covering for dermal ulcers and defects. It is designated as a Human Cell & Tissue Product (HCT/P) by the U.S. FDA.

DETAILED DESCRIPTION:
Patients identified for the study will have a non-healing diabetic ulcer, between 1-25cm² in size. The patient's wound(s) will be monitored for 2 weeks to document the wound pathology. Patients with less than 30% wound area reduction during the 2 week screening period and who meet all of the inclusion and none of the exclusion criteria, will be enrolled in the study. All patients will be assigned to a study or control group and undergo sharp debridement. NEOX® CORD 1K matrix will be applied to the treatment group on the day of debridement, covered with a wound veil, and standard dressing. Both groups will be monitored weekly, and the % decrease in wound size will be recorded at Baseline and Weeks 1, 2, 3, 4, 6, 8 and 12. If the wound is not progressing, additional application of NEOX® CORD 1K may be applied. The time to complete closure will be recorded for both groups. The study duration will be 12 weeks. Subjects in the control group that continue to suffer a non-healing wound at the week 12 visit will be offered an opportunity to cross-over to NEOX treatment and followed for an additional 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 years and 80 years of age inclusive
2. Confirmed diagnosis of Type I or Type II Diabetes
3. Males and Females diagnosed with a diabetic foot ulcer that is 1-25cm²
4. At least one foot ulcer that is UT Grade IA
5. Evidence of proper circulation which includes: An Index Ulcer defined as chronic (presence of wound for > 4 weeks) but not present for more than 52 weeks at the Screening Visit
6. The Index Ulcer is located below the malleoli on the plantar or dorsal surface of the foot
7. The Index Ulcer extends into the dermis or subcutaneous tissue with no evidence of exposed muscle, tendon, bone, or joint capsule
8. Wound is free of necrotic debris and clinical signs of infection
9. Patient has adequate circulation to the foot
10. In patients with non-compressible ankle vessels there is adequate flow to the foot.

Exclusion Criteria:

1. The Index Ulcer is of non-diabetic pathophysiology and/or over an active Charcot deformity
2. The Index Ulcer is UT Grade IB or higher (worsening)
3. Gangrene is present on any part of the affected foot
4. The longest dimension of the Index Ulcer exceeds 5 cm at the Baseline Visit
5. Patient is currently receiving renal dialysis
6. Patient has a glycated hemoglobin A1c (HbA1c) level of > 12%
7. Patient has significant renal impairment
8. Chronic oral steroid use > 7.5 mg daily
9. Requiring intravenous (IV) antibiotics to treat the index wound infection
10. Patient has an ulcer within 15cm of the Index Ulcer identified for study consideration
11. Patient is receiving oral or parenteral corticosteroids, immunosuppressive or cytotoxic agents
12. Patient is Human Immunodeficiency Virus (HIV) positive or has Acquired Immune Deficiency Syndrome (AIDS)
13. Current evidence of osteomyelitis, cellulitis, or other evidence of infection including fever or purulent drainage from the wound site
14. Patient has active malignancy other than non-melanoma skin cancer
15. Patient's Index Ulcer has decreased by ≥ 30% during 2-week screening period
16. Patient has untreated alcohol or substance abuse at the time of screening
17. Pregnant women
18. Patient is currently enrolled or participated in another investigational device, drug, or biologic trial within 60 days of screening
19. Patient has allergy to primary or secondary dressing materials used in this trial
20. Patient has an allergy to amphotericin-B or Dulbecco's Modified Eagle Medium (DMEM)
21. Patient has had within the last 30 days, or is currently undergoing, or is planning for wound treatments with enzymes, growth factors, living skin, dermal substitutes or other advanced biological therapies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Complete wound closure | 12 weeks
  Complete closure of the index wound, defined as 100% re-epithelialization as determined by the Investigator
Number of participants with adverse events | 12 weeks
  Number of participants with adverse events will be compared between the two groups.

SECONDARY OUTCOMES:
Number of applications | 12 weeks
  Number of applications of study product (up to 12 weeks from Baseline)
Blinded Reader Assessment | 12 weeks and 24 weeks
  Percent of wounds achieving complete closure per the assessment of a Blinded Reader (by blinded photograph of wound and measurement acetate).
Time to Initial Wound Closure | Up to 12 weeks or 24 weeks (Crossover)
  Time to initial wound closure (Up to12 weeks from Baseline or 24 weeks for crossover group)

CONTACTS AND LOCATIONS:
Overall Officials: Charles I. Romano, Study Director — Amniox Medical, Inc.
Locations (3):
- United States (3):
  - University of Arizona, Tucson, Arizona
  - Center for Clinical Research, Inc., Castro Valley, California
  - Ankle and Foot Centers of Georgia, Newnan, Georgia